CLINICAL TRIAL: NCT07304362
Title: The Effect of Education Given to School-Age Children With Cystic Fibrosis and Their Parents on Health Literacy Levels
Brief Title: The School-Age Children With Cystic Fibrosis and Their Parents on Health Literacy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Duygu Demir, PhD, RN, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: duygudemir KF Burcu
Record Dates: First submitted 2025-11-28; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Cystic Fibrosis (CF)
Keywords: cystic fibrosis; Health Literacy; Chronic Disease; School-Age Child
MeSH Terms: conditions — Cystic Fibrosis; Chronic Disease

STUDY DESIGN:
Intervention Model Description: The study is planned to be conducted as a randomized controlled experimental design with a pretest-posttest structure. The research will consist of two groups: an intervention group receiving the online education program and a control group receiving no additional intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Education Group (Experimental)
  Interventions: Behavioral: Online Education Program
- Control Group (No Intervention): Children in the control group will receive only routine follow-up and standard care. No additional intervention will be provided to this group.

INTERVENTIONS:
Behavioral: Online Education Program — Children with cystic fibrosis and their parents in the intervention group will receive an online education program designed to improve health literacy. The program will be delivered once, immediately after the pretest, through an online platform. The session will last approximately 30-40 minutes and will follow a standardized educational protocol reviewed by expert faculty members. Posttest assessment will be conducted 4 weeks after the intervention. The program aims to enhance parents' ability to interpret, apply, and make decisions based on health information, and to help children understand and take responsibility for their own health.
  Arms: Online Education Group

SUMMARY:
This randomized controlled experimental study is planned to examine the effect of an online education program provided to school-age children aged 6-11 years diagnosed with cystic fibrosis and their parents on health literacy levels.

The study population will consist of 123 school-age children with cystic fibrosis and their parents who are followed at the Cystic Fibrosis Outpatient Clinic of Marmara University Pendik Training and Research Hospital. The study sample will include 104 children and their parents, who will be randomly assigned to either the intervention group (n = 52) or the control group (n = 52).

Data will be collected using the Introductory Information Form, the Health Literacy Scale for School-Age Children, and the Turkey Health Literacy Scale-32. Following the pre-test assessments, an online education program developed by the researcher will be delivered to the intervention group. The control group will not receive any additional intervention. Both groups will complete post-test assessments four weeks after the pre-test.

DETAILED DESCRIPTION:
The study population will consist of school-age children aged 6-11 years who are diagnosed with cystic fibrosis and meet the inclusion criteria, along with their parents, followed at the Cystic Fibrosis Outpatient Clinic of Marmara University Pendik Training and Research Hospital.

This study is planned to be designed as a randomized controlled experimental study with a pretest-posttest design in order to determine the effect of an online education program that will be delivered to children with cystic fibrosis and their parents on health literacy levels. The study will aim to evaluate parents' ability to understand, evaluate, and use health information accurately, as well as children's understanding of their disease, their responsibility in managing their health, and the development of healthy lifestyle behaviors.

To ensure homogeneous distribution of the groups, randomization will be performed using a computer-based system (http://www.randomization.com, balanced permutation method). Children who meet the inclusion criteria and whose parents provide consent will be randomly assigned to either the intervention group or the control group according to the randomization list.

The online education program, developed by the researcher, will be administered to the intervention group following the pretest. The control group will not receive any additional intervention. Both groups will complete posttest assessments four weeks after the pretest.

Study Variables

• Independent Variable: The independent variable of the study will be the online education program that will be delivered to school-age children with cystic fibrosis and their parents.

• Dependent Variables: The dependent variables will be the health literacy levels of children diagnosed with cystic fibrosis and their parents.

• Control Variables: The control variables will include the descriptive characteristics of the children (age, gender).

ELIGIBILITY:
Inclusion Criteria:

Children aged 6-11 years at the time of the study.

Children receiving treatment at the Cystic Fibrosis Diagnosis and Treatment Center during the study period.

Children able to understand and complete the Health Literacy Scales (no visual, auditory, or cognitive impairments that would prevent scale completion).

Children with sufficient proficiency in Turkish to answer the scales.

Children and parents who voluntarily agree to participate.

Children who have not previously received any health literacy education.

Exclusion Criteria:

Children with severe visual, auditory, or cognitive impairments that would prevent them from understanding or completing the scales.

Children who have already received health literacy education.

Children who are outside the age range of 6-11 years.

Children not receiving follow-up at the Cystic Fibrosis Diagnosis and Treatment Center during the study period.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Children's health literacy levels | 4 weeks after the intervention
  Will be assessed using the Health Literacy Scale for School-Age Children, indicating the child's ability to understand, interpret, and apply health information.
Parents' health literacy levels | 4 weeks after the intervention
  Will be measured via the Turkey Health Literacy Scale-32 to assess parents' ability to understand, interpret, and apply health-related information.

CONTACTS AND LOCATIONS:
Locations (1):
- Yalova Universty, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cordeiro SM, da Silva HB, Silva-Rodrigues FM. Family caregivers' needs for information on pediatric cystic fibrosis: A qualitative study. J Child Health Care. 2024 Nov 26:13674935241303539. doi: 10.1177/13674935241303539. Online ahead of print. PMID 39589857
- [Background] Yuksek BN, Ayaz-Alkaya S. Effectiveness of health literacy education on health literacy in early adolescence: A randomized controlled trial. Public Health. 2024 Dec;237:135-140. doi: 10.1016/j.puhe.2024.09.024. Epub 2024 Oct 9. PMID 39383558
- [Background] Ahmadpour M, Omidvar N, Shakibazadeh E, Doustmohammadian A, Rahimiforoushani A. Development and evaluation of an intervention to improve food and nutrition literacy among Iranian Kurdish primary school children: An application of intervention mapping approach. Front Public Health. 2023 Jan 4;10:1059677. doi: 10.3389/fpubh.2022.1059677. eCollection 2022. PMID 36684859
- [Background] McDonald CM, Haberman D, Brown N. Self-efficacy: empowering parents of children with cystic fibrosis. J Cyst Fibros. 2013 Sep;12(5):538-43. doi: 10.1016/j.jcf.2012.11.014. Epub 2012 Dec 24. PMID 23269367
- [Result] de Buhr E, Tannen A. Parental health literacy and health knowledge, behaviours and outcomes in children: a cross-sectional survey. BMC Public Health. 2020 Jul 13;20(1):1096. doi: 10.1186/s12889-020-08881-5. PMID 32660459
- [Result] Li Y, Xiao Q, Chen M, Jiang C, Kang S, Zhang Y, Huang J, Yang Y, Li M, Jiang H. Improving Parental Health Literacy in Primary Caregivers of 0- to 3-Year-Old Children Through a WeChat Official Account: Cluster Randomized Controlled Trial. JMIR Public Health Surveill. 2024 Jul 4;10:e54623. doi: 10.2196/54623. PMID 38989817
- [Result] Broder J, Okan O, Bauer U, Bruland D, Schlupp S, Bollweg TM, Saboga-Nunes L, Bond E, Sorensen K, Bitzer EM, Jordan S, Domanska O, Firnges C, Carvalho GS, Bittlingmayer UH, Levin-Zamir D, Pelikan J, Sahrai D, Lenz A, Wahl P, Thomas M, Kessl F, Pinheiro P. Health literacy in childhood and youth: a systematic review of definitions and models. BMC Public Health. 2017 Apr 26;17(1):361. doi: 10.1186/s12889-017-4267-y. PMID 28441934